CLINICAL TRIAL: NCT05469308
Title: Predictivity and Evaluation of the Adherence of Ambulatory Patients Treated With a Direct Oral Anticoagulant for Atrial Fibrillation
Brief Title: Adherence to Oral Anticoagulants in Patients With Atrial Fibrillation
Acronym: 3AOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0020
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-06

CONDITIONS: Oral Anticoagulant; Adherence
Keywords: Direct oral anticoagulant; Adherence; Proportion of days covered; adherence questionary; Girerd adherence questionary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- questionary (Experimental)
  Interventions: Other: questionary

INTERVENTIONS:
Other: questionary — When the patients renew their treatment in community pharmacy, they have an adherence record with a pharmacist who calculates the PDC score, and perform questionaries on adherence to the DOACs, and collects data about clinical history and pharmacological information on the prescribed DAOCs, demography.

SUMMARY:
The rhythm disorders of Atrial Fibrillation (AF) require continuous treatment with anticoagulants to prevent stroke. The introduction of direct oral anticoagulants (DOACs) quickly supplanted the administration of anti-vitamin K (AVK) which presented an elevated risk of hemorrhage.

However, the adherence of the treatments by the OAD is very poor, several studies show that 30 to 50% of the patients fail to adhere to their treatment very soon after starting it. In a recent study, in the United States, using data collected between 2010 and 2014 in more than 60,000 patients with AF, Yao et al show that less than 50% of patients can be considered "adherent".

They conclude in this study that adherence to anticoagulation is low in practice, although it may be slightly improved with DOACs. More recently a meta-analysis shows that 66% of patient treated by DOACs were considered adherent (PDC > 80 %). In addition, therapeutic adherence seems to be essential in patients with a CHA2DS2-VASc score ≥2. Indeed improving adherence reduces the risk of stroke occurrence. The investigators propose to evaluate during an interview in the pharmacy, the adherence of ambulatory patients (at the time of their renewal of treatment at the pharmacy) by the "Proportion of Days Covered" (PDC) of the treatment by AOD, and by a simplified questionnaire and to define a profile of patients treated for AF at risk of nonadherence to AOD (PDC adherence prediction score). The investigators perform an observational, prospective multicenter study , in which patients adherence will be quantified in a standardized method.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Consultation in the community pharmacy
* long-term treatment for at least six months with an DOACs.
* Patients able and agreeing to participate in the evaluation of their adherence

Exclusion Criteria:

* Treatment by DOACs limited in the duration
* Contra-indications of DOACs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Number of AOD specific PDC | 2 years
  Determination of the AOD (Direct oral anticoagulants) specific PDC (Proportion of Days Covered) of patients coming to renew their treatment in the community pharmacy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No